CLINICAL TRIAL: NCT06578091
Title: Effects of Executive Dysfunction on Physical Performance and General Well-Being in Obese Individuals
Brief Title: Executive Function in Obese
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Okur, Assist. Prof., Kutahya Health Sciences University
Other Study IDs: KSBU-2024/03-33
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: obesity; executive functions; physical performance; well-being
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Executive Function Deficit Group
- Control Group

SUMMARY:
This study was planned to examine the effect of executive function problems on physical performance and general well-being in obese individuals.

ELIGIBILITY:
Inclusion Criteria:

For the study group;

* Individuals volunteering for the study with BMI ≥30 kg/m2
* Individuals between the ages of 18-65 who volunteer to work
* Individuals who scored 21 points and above in the cognitive assessment

For the control group;

* Individuals volunteering for the study with BMI ≥30 kg/m2
* Individuals between the ages of 18 and 65 who are willing to work
* Scoring less than 21 points on the cognitive assessment

Exclusion Criteria:

* Being at a mental level that cannot understand and answer the questions posed
* Having a diagnosed neurological disease
* Having had cancer within the last 2 years
* Having major organ dysfunction
* Having uncontrolled type 2 diabetes
* Loss of vision, hearing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with BMI ≥30 kg/m2
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Executive function | Baseline
  It will be assessed with the Montreal Cognitive Assessment. Accordingly, a score of 21 points and above is considered normal. Individuals who score 21 points or less on this test will be included in the executive function deficit group. The others will included in control group.
General Well-Being-Sleep Quality | Baseline
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index. The scale consists of 18 questions and 7 components and was developed to assess sleep disturbances and sleep quality in the last 1 month. These components include subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleep medication use and daytime dysfunction. For scoring, it is applied as 0 if it has never occurred during the last month, 1 if it occurs less than once a week, 2 if it occurs once or twice a week, and 3 if it occurs three or more times a week. The total score has a value between 0-21. If the total score obtained as a result of the questionnaire is above 5, sleep quality is clinically poor.
General Well-Being-Quality of Life | Baseline
  Quality of life, sleep quality and depression levels will be assessed. Quality of life will be assessed with the 12-item Short Health Scale. Short Health Scale consists of 8 sub-dimensions and 12 items including physical functioning (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functioning (1 item), emotional role (2 items) and mental health (2 items). Items related to physical and emotional role are answered as yes or no, while other items have Likert-type options ranging from 3 to 6. A higher score represents better health.
Physical Performance-Timed Up and Go | Baseline
  The timed up and go test is a functional dynamic balance test. The Timed Up and Go test is a timed measurement in which the individual has to get up from a chair, walk 3 meters, turn around, walk back and sit down. The Timed Up and Go is used to assess functional mobility and dynamic balance control in older people to identify increased risk of falls. Participants will be asked to wear the shoes they regularly wear to walk at a normal pace and will be allowed walking aids. The time between the participants getting up from the chair and sitting down again will be recorded in seconds.
General Well-Being-Depression and Anxiety | Baseline
  Depression and anxiety level will be assessed with the Hospital Depression and Anxiety Scale. It consists of 14 items. Seven of these items measure anxiety and the other seven items measure depression symptoms. The items in the scale are evaluated with a 4-point Likert scale and are based on a scoring system between 0-3. According to the scoring, 0-1 is considered as not ill, 2 as borderline ill, and 2-3 as severely ill. Higher scores indicate more severe depression and anxiety.
Physical Performance-Hand Grip Strength | Baseline
  A digital Jamar dynamometer calibrated for hand grip strength (Performance Health, Warrenville, IL), Participants will be instructed to squeeze the dynamometer as hard as possible while sitting in an upright position as recommended by the American Association of Hand Therapists, with arms at their sides, elbows flexed 90° and forearms in a neutral position. A trial will be requested beforehand. For hand grip strength, 3 measurements will be made with one-minute intervals between each measurement and the average value will be recorded.
Physical Performance-Walking Speed | Baseline
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. A clear distance of at least 10 meters in length will be determined and marks will be added at 2 meters and 8 meters. Timing will start when the individual's toes cross the 2 meter mark. The person will be instructed to walk as fast as you can safely walk until I say stop. The timing will stop when the toes cross the 8 meter mark. Three trials will be performed and the average of the three trials will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No